CLINICAL TRIAL: NCT06798337
Title: The Effect of Reward on Cognitive Functioning, Motor Skills, and Motivation in 8- to 10-Year-Old Children With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Reward Effects on Cognition, Motor Skills, and Motivation in Children
Acronym: ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Principal Investigator, Vilma Dudoniene, assoc. prof. dr., Lithuanian Sports University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Lithuanian Sports University
Record Dates: First submitted 2025-01-15; First posted 2025-01-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Attention-Deficit/Hyperactivity Disorder (ADHD)
Keywords: attention; motor skills; motivation; reward-based therapy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Qualitative research
Who Masked: Participant, Investigator
Masking Description: Reword group did not know about conventional PT group and vice versa.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional outpatient PT group (n=30). (Experimental): Conventional outpatient PT group received typical physical exercises with duration of 6 weeks
  Interventions: Other: Conventional Physiotherapy group
- Reward-based PT group (Experimental): This group received reward based virtual reality exercises with duration of 6 weeks. Reward was extra exercises using virtual reality
  Interventions: Other: Reward based physiotherapy group

INTERVENTIONS:
Other: Conventional Physiotherapy group — Participants in the regular physical therapy group performed balance and coordination exercises three times a week without the use of rewards. These subjects completed only physical exercises, without engaging in game-like interactive tasks using virtual reality (VR) glasses. Each session was conducted at the same time for each subject, with a potential variation of ±1 hour.
  Arms: Conventional outpatient PT group (n=30).
Other: Reward based physiotherapy group — Subjects in the reward group performed balance and coordination exercises three times a week, with the inclusion of rewards. At the end of each exercise session, participants engaged in game-like interactive tasks using virtual reality (VR) glasses. Exercise sessions were conducted at the same time for each subject, with a permissible variation of ±1 hour.
  Arms: Reward-based PT group

SUMMARY:
This interventional study aimed to aimed to evaluate the effects of rewards on cognitive function, motor skills, and motivation in 8- to 10-year-old children with ADHD following 3- and 6-week interventions.

DETAILED DESCRIPTION:
Research problem: children with Attention-Deficit/Hyperactivity Disorder (ADHD) are inattentive and distractible, which often makes it difficult for physiotherapists to keep them interested, as prolonged activity often causes boredom.

The aim of this study was to determine the effects of reward on cognitive function, motor skills and motivation in 8-10 year old children with ADHD after 3 and 6 week interventions.

Objectives of the study:

1. To compare the cognitive function of children receiving conventional physiotherapy with that of children receiving reward therapy. 2. To compare the motor skills of the children receiving conventional physiotherapy with those of the children receiving the reward. 3. To compare the motivation of children receiving conventional physiotherapy with that of children receiving rewards.

The hypothesis of the study is that exercise with rewards improves cognitive function, motor skills and motivation better than conventional physiotherapy in children aged 8 to 10 years with attention deficit disorder.

Research methods: the study included 60 boys diagnosed with ADHD. Age: 8-10 years. Subjects were randomly divided into reward and conventional physiotherapy groups. In both groups, subjects performed exercises for balance and coordination for 3 times per week for 45 min, but in one group subjects received a reward using virtual reality.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ADHD confirmed by a neurologist;
2. male gender;
3. age between 8 and 10 years.
4. ability to read and write;
5. patient's willingness to attend physiotherapy sessions;

Exclusion Criteria:

1. claustrophobia;
2. neurological disorders (e.g., autism spectrum disorder, depression, obsessive-compulsive disorder, Tourette's syndrome);
3. chronic medical conditions (e.g., cancer, diabetes, cardiovascular diseases);
4. previous treatment for ADHD (e.g., pharmacological therapy, cognitive behavioral therapy) within the last six months;
5. Medication use.

Ages: 8 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Boys were invited to participate in the study.
Enrollment: 67 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Static balance | At baseline and after 6 weeks
  was assessed with The Abili Balance Analyzer platform. The software associated with the platform provided an overall stability index based on the tests conducted: Very Good: 0.8; Good: 0.8 to 1.8; Poor: >1.8.
Attention task with spatial numbers | At baseline and after 6 weeks
  Number of mistakes and Speed coefficient was recorded.
Attention task with spatial figures | At baseline and after 6 weeks
  Number of mistakes and Speed coefficient was recorded.
Easy figural memory task | At baseline and after 6 weeks
  Number of mistakes and Speed coefficient was recorded.
Hard figural memory task | At baseline and after 6 weeks
  Number of mistakes and Speed coefficient was recorded.
Visuo-Constructional Ability task | At baseline and after 6 weeks
  Number of successful attempts and duration (in seconds) was recorded

SECONDARY OUTCOMES:
Pediatric motivation Scale (PMot) | At baseline and after 6 weeks
  Participants were instructed to respond to the questions by selecting a visual image that best represented their emotional state. Each visual image was assigned a numerical value, ranging from 1 (very poor) to 6 (excellent), for statistical data analysis and outcome evaluation (numeric value).

CONTACTS AND LOCATIONS:
Overall Officials: Vilma VD Dudoniene, PhD, Principal Investigator — Lithuanian Sports University; Vilma Dudoniene, PhD, Study Chair — Lithuanian Sports University
Locations (1):
- Department of health promotion and rehabilitation, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No
The consent form of the informed person states that the individual data of the subjects will not be disclosed, but can only be used to summarized.